CLINICAL TRIAL: NCT01662076
Title: A Feasibility Pilot Trial of Individualized Homeopathic Treatment of Fatigue in Children Receiving Chemotherapy
Brief Title: Homeopathic Treatment of Fatigue in Children Receiving Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lillian Sung, Staff Physician, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1000027444
Record Dates: First submitted 2012-08-02; First posted 2012-08-10 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Cancer
Keywords: Cancer; Fatigue; Chemotherapy; Pediatrics; Homeopathy
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Materia Medica

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sublingual or Oral Liquid Homeopathy (Experimental): The homeopathic remedy will be administered as 1 lactose/sucrose globule 2.5 mm in diameter to be administered sublingually up to 3 times per day or as 0.2 ml of a 30% ethanol based liquid homeopathic remedy administered orally up to 3 times per day. The homeopathic remedy and/or the homeopathic remedy potency can be changed on a daily basis during the course of treatment. However, only one homeopathic remedy and potency will be administered at a given time.
  Interventions: Other: Homeopathic Remedies

INTERVENTIONS:
Other: Homeopathic Remedies — The homeopathic remedy will be administered as either 1 globule sublingual or 0.2 mL oral (depending on chosen formulation) up to 3 times per day. The homeopath will decide which formulation will be used. Homeopathic remedies prepared according to the standards as set out by Health Canada. The caregiver or patient will be asked to administer the homeopathic remedy at least 30 minutes before or after taking other medications, food and strong smelling substances (such as camphor, mint, or coffee).

SUMMARY:
Cancer-related fatigue has been described as a subjective feeling of physical, emotional, and/or cognitive tiredness. Fatigue is frequently identified as one of the most troublesome symptoms in pediatric cancer patients. Fatigue affects children with cancer throughout the trajectory of their disease. Treatment interventions for cancer-related fatigue have been largely unsuccessful. Homeopathy involves treatment of patients with diluted natural substances aimed at stimulating the body's healing system. In the efficacy trial literature, individualized homeopathy shows the most promise over other forms of homeopathic intervention. Individualized homeopathic treatment involves a unique yet established method of case taking. During the consultation, the homeopath asks a series of broad questions to elicit subjective symptoms related to the patient's disease, their medical history, as well as particular characteristics (physical or psychological) related to the individual. This study will recruit children receiving chemotherapy to undergo homeopathic remedies to treat their fatigue. This study hypothesizes that homeopathic treatment will effectively treat fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with any type of cancer. Patients may have newly diagnosed, relapsed or a second malignant disease.
* Receiving any type of chemotherapy administered intermittently (i.e. not continuous administration) with or without radiation treatment
* Discharge from SickKids is anticipated to occur following completion of the current inpatient chemotherapy or chemotherapy is being administered as an outpatient
* Between 2 and 18 years of age (age range for which instruments are available and children may be able to comply with homeopathy) A score on the Symptoms Distress Scale (SDS) of 2 or higher
* Able to ingest medications in lactose/sucrose globule or liquid form
* Reside within Greater Toronto area or willing to travel to the Riverdale Homeopathic Clinic. Participants living outside of the Greater Toronto area who wish to receive home visits may be eligible provided that permission is granted by the homeopath investigator
* A parent or caregiver must be able to read and write in English.
* Patients who are currently receiving CAM including homeopathy are eligible.

Exclusion Criteria:

* Previous history of allergy to the homeopathic products

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2012-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | baseline
  The primary objective is to determine the feasibility of recruiting patients for a study of individualized homeopathy in paediatric patients receiving chemotherapy for cancer.

SECONDARY OUTCOMES:
Feasibility of administration | 14 days
  To determine the feasibility of administering individualized homeopathy in pediatric cancer patients receiving chemotherapy for cancer by describing the proportion of participants who complete at least 10 days of treatment
Changes in fatigue | Change from baseline to 14 days
  To describe changes in fatigue scores according to the Symptom Distress Scale (SDS) and the PedsQL Multidimension Fatigue Scale
Changes in quality of life | Change from baseline to 14 days
  To describe changes in generic and cancer specific quality of life as measured by the PedsQL Generic Core Scales and Acute Cancer Module

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Sung, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada